CLINICAL TRIAL: NCT03487562
Title: A Randomized, Open-label, Multiple Dose, Two-part Phase I Clinical Trial to Compare the Pharmacokinetics, Pharmacodynamics and Safety/Tolerability of DWP14012 After Administrations of DWP14012 Alone and Combinations of DWP14012, Clarithromycin and Amoxicillin in Healthy Male Subjects
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of After Administrations of DWP14012 Alone and Combinations of DWP14012, Clarithromycin and Amoxicillin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWP14012003
Record Dates: First submitted 2018-03-13; First posted 2018-04-04 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Healthy
MeSH Terms: interventions — Clarithromycin; Amoxicillin; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Sequence 1 (Experimental): Part I: A-B-D-C A: DWP14012 A mg bid B: DWP14012 A mg bid + Clarithromycin 500 mg bid C: DWP14012 A mg bid + Clarithromycin 500 mg bid + Amoxicillin 1 g bid D: Clarithromycin 500 mg bid + Amoxicillin 1 g bid
  Interventions: Drug: DWP14012 Amg; Drug: Clarithromycin; Drug: Amoxicillin
- Sequence 2 (Experimental): Part I: B-C-A-D A: DWP14012 A mg bid B: DWP14012 A mg bid + Clarithromycin 500 mg bid C: DWP14012 A mg bid + Clarithromycin 500 mg bid + Amoxicillin 1 g bid D: Clarithromycin 500 mg bid + Amoxicillin 1 g bid
  Interventions: Drug: DWP14012 Amg; Drug: Clarithromycin; Drug: Amoxicillin
- Sequence 3 (Experimental): Part I: C-D-B-A A: DWP14012 A mg bid B: DWP14012 A mg bid + Clarithromycin 500 mg bid C: DWP14012 A mg bid + Clarithromycin 500 mg bid + Amoxicillin 1 g bid D: Clarithromycin 500 mg bid + Amoxicillin 1 g bid
  Interventions: Drug: DWP14012 Amg; Drug: Clarithromycin; Drug: Amoxicillin
- Sequence 4 (Experimental): Part I: D-A-C-B A: DWP14012 A mg bid B: DWP14012 A mg bid + Clarithromycin 500 mg bid C: DWP14012 A mg bid + Clarithromycin 500 mg bid + Amoxicillin 1 g bid D: Clarithromycin 500 mg bid + Amoxicillin 1 g bid
  Interventions: Drug: DWP14012 Amg; Drug: Clarithromycin; Drug: Amoxicillin
- A (Experimental): Part II: (DWP14012 B mg + Clarithromycin 500 mg + Amoxicillin 1g) bid
  Interventions: Drug: DWP14012 Bmg; Drug: Clarithromycin; Drug: Amoxicillin
- B (Experimental): Part II: (DWP14012 A mg + Clarithromycin 500 mg + Amoxicillin 1g) bid
  Interventions: Drug: DWP14012 Amg; Drug: Clarithromycin; Drug: Amoxicillin
- C (Experimental): Part II: (Lansoprazole 30 mg + Clarithromycin 500 mg + Amoxicillin 1g) bid
  Interventions: Drug: Clarithromycin; Drug: Amoxicillin; Drug: Lansoprazole

INTERVENTIONS:
Drug: DWP14012 Amg — DWP14012 Amg
  Arms: B; Sequence 1; Sequence 2; Sequence 3; Sequence 4
Drug: DWP14012 Bmg — DWP14012 Bmg
  Arms: A
Drug: Clarithromycin — Clarithromycin 500 mg
Drug: Amoxicillin — Amoxicillin 1 g
Drug: Lansoprazole — Lansoprazole 30 mg
  Arms: C

SUMMARY:
This is a randomized, open-label, multiple dose, two-part phase I clinical trial to compare the pharmacokinetics, pharmacodynamics and safety/tolerability of DWP14012 after administrations of DWP14012 alone and combinations of DWP14012, Clarithromycin and Amoxicillin in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged between 19 and 50 at screening
* Those whose weight is between 55 and 90 kg and BMI is between 18.0 and 27.0
* Part I: Those who have been helicobacter pylori negative at screening Part II: Those who have been helicobacter pylori positive at screening
* Those who are adequate to be subjects in this study upon judgment of the investigator after physical examination, clinical laboratory test, examination by interview, etc

Exclusion Criteria:

* Those who have clinical significant liver, kidney, nervous system, respiratory, endocrine, hematology and oncology, cardiovascular, urinary, and mental diseases or past history
* Those who have gastrointestinal diseases or past history of gastrointestinal diseases (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux, Crohn's disease etc.) that may affect safety and pharmacokinetic/pharmacodynamic evaluation of study drug, and those who have past history of gastrointestinal surgery (however, except simple appendectomy and herniotomy)
* Those whose plasma AST (SGOT) and ALT (SGPT) exceed to the upper limit of the normal range
* Those who have anatomical disability in insertion and maintenance of pH meter catheter

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Cmax,ss: Maximum concentration of DWP14012, clarithromycin and metabolite and amoxicillin at steady state | Day 1~7 pre-dose, Day 8 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Part I: each period (Group A, B, C, D) Part II: Group A, B
Cmin,ss: Minimum concentration of DWP14012, clarithromycin and metabolite and amoxicillin at steady state | Day 1~7 pre-dose, Day 8 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Part I: each period (Group A, B, C, D) Part II: Group A, B
Cav,ss: Average concentration of DWP14012, clarithromycin and metabolite and amoxicillin at steady state | Day 1~7 pre-dose, Day 8 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Part I: each period (Group A, B, C, D) Part II: Group A, B
AUCt,ss: Area under the drug concentration-time curve within a dosing interval at steady states | Day 1~7 pre-dose, Day 8 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Part I: each period (Group A, B, C, D) Part II: Group A, B
Tmax,ss: Time of maximum concentration at steady state | Day 1~7 pre-dose, Day 8 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Part I: each period (Group A, B, C, D) Part II: Group A, B
T1/2: Elimination half-life | Day 1~7 pre-dose, Day 8 pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 hours
  Part I: each period (Group A, B, C, D) Part II: Group A, B
Percentage of total time that the intragastric pH was above 4 | Period 1 Day -1 and Group A, C Day 7 0~24 hours
  Part I
Percentage of total time that the intragastric pH was above 4 | Day -1, Day 1, Day 7 0~24 hours
  Part II
Percentage of total time that the intragastric pH was above 6 | Period 1 day -1 and Group A, C Day 7 0~24 hours
  Part I
Percentage of total time that the intragastric pH was above 6 | Day -1, Day 1, Day 7 0~24 hours
  Part II
Serum gastrin concentration profile | Period 1 Day -1 and Group A, C Day 7 pre-dose, 2, 4, 6, 8, 12, 24, 48 hours
  Part I
Serum gastrin concentration profile | Day -1 pre-dose, 2, 4, 6, 8, 12 hours, Day 1 and 7 pre-dose, 2, 4, 6, 8, 12, 24, 48 hours
  Part II
Number of participants with Adverse Events (AE) | Day -2 (Randomization) to Day 60 (Post-study visit of Part I) and Day 42 (Follow up visit of Part II)
  All AE standardized using MedDRA was assessed by investigator using the protocol defined grading system. Intensity was categorized as mild, moderate and severe
Number of Participants With Clinically Significant Vital Sign findings | Day -2 (Randomization) to Day 60 (Post-study visit of Part I) and Day 42 (Follow up visit of Part II)
  Blood pressure(mmHg), pulse (beats/min) and body temperature(℃) were tested. The Average, Median, Standard Deviation, Min, Max values will be calculated to assess the safety/tolerability.
Number of Participants With Clinically Significant Electrocardiogram(12-lead ECG) findings | Day -2 (Randomization) to Day 54~60 (Post-study visit of Part I) and Day 36~42 (Follow up visit of Part II)
  Ventricular rate(beats/min), RR, PR interval(msec), QRS duration(msec), QTcB and QTcF were recorded. The results of 12-lead ECG will be categorized Normal/Abnormal NCS(No clinically significant)/Abnormal CS(clinically significant).
Number of Participants With Clinically Significant Laboratory results | Day -2 (Randomization) to Day 60 (Post-study visit of Part I) and Day 42 (Follow up visit of Part II)
  Hematology, Blood chemistry, Coagulation and Urinalysis were tested. The Average, Median, Standard Deviation, Min, Max values will be calculated to assess the safety/tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea